CLINICAL TRIAL: NCT01725204
Title: A Safety and Efficacy Study of Adding Low Dose Pegylated IFN-alpha 2B to Standard Dose Dasatinib in Patients With Newly Diagnosed Chronic Phase Myeloid Leukemia
Brief Title: Safety and Efficacy of Pegylated IFN-alpha 2B Added to Dasatinib in Newly Diagnosed Chronic Phase Myeloid Leukemia
Acronym: NordCML007
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NordCML007; 2011-005989-38 (EudraCT Number)
Record Dates: First submitted 2012-11-08; First posted 2012-11-12 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2017-09

CONDITIONS: Leukemia, Myeloid, Chronic-Phase
Keywords: dasatinib; Protein Kinase Inhibitors; pegylated IFN-alpha 2B; Interferon-alpha
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase | interventions — Dasatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dasatinib + PegIFN (Experimental): Dasatinib 100mg OD for three months single drug, with subsequent addition of PegIFN 15 μg/ week for 3 months. If well tolerated (less than grade 2 non-hematological or grade 3 hematological AE) the dose should be increased to 25μg weekly for the remaining 9 months on combination treatment. Thereafter dasatinib will be given as monotherapy. Patients will be followed for 24 months totally.
  Interventions: Drug: Dasatinib + PegIFN

INTERVENTIONS:
Drug: Dasatinib + PegIFN

SUMMARY:
Patients with newly diagnosed CML have excellent outcomes with tyrosine kinase inhibitors (TKI). However, a few patients will be cured with TKIs alone, and thus need continued life-long treatment. Some patients achieve complete molecular remission (CMR), and this rate is higher with second generation TKIs compared with imatinib. Some experience with drug discontinuation in CMR has been derived from a few small studies, most notably the French STIM study. Approximately 40 % of patients with a minimum of two years in MR4.5 (4.5 log reduction in molecular response) can stop imatinib without relapse, indicating possible cure. To increase the non-relapse rate is of major importance. To achieve a permanent "cure" without stem cell transplantation is presently the most relevant goal of clinical studies in CML.

The investigators hypothesize that to significantly increase cure rates in CML, therapy should eradicate leukemic stem cells and/or induce or restore anti-CML immunity. Second generation TKIs may have a more profound effect on the stem cell pool as compared to imatinib. This is assessed in our current randomized study with a reduction in leukemic stem cell burden as the primary endpoint (NordCML006). Interferon-alpha (IFN) has a prominent immunomodulatory and antiproliferative mode of action, and has also activity in stem cells. Pegylated IFN in combination with imatinib results in improved therapy responses as compared to imatinib monotherapy. This advantage may translate into higher cure rates.

Dasatinib has a unique dual mechanism of action: it is the most potent of available TKIs and induces immunological effects that are different from those of IFN. Both of these drugs may have immunological adverse-effects when used as a monotherapy. However, immunological adverse-effects may also be markers of anti-leukemia efficacy. A combination of dasatinib and pegylated IFN (PegIFN) may have additive or synergistic effects and should be tested in a clinical study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of chronic myeloid leukemia in chronic phase (CML-CP) associated with BCR-ABL1 quantifiable by RQ-PCR (IS)
* No other current or planned anti-leukemia therapies excluding hydroxyurea treatment for up to two months.
* ECOG Performance status 0,1, or 2
* Adequate organ function as defined by: Total bilirubin < 1.5 x ULN (ULN = upper limit of normal in a local institution lab) in absence of Gilbert genotype; ASAT and ALAT < 2.5 x ULN. Creatinine < 2x ULN. Potassium, magnesium and phosphate not below LLN (LLN= lower level of normal)
* Life expectancy of more than 12 months in the absence of any intervention
* Patient has given written informed consent to participate in the study

Exclusion Criteria:

* Prior accelerated phase or blast crisis
* Uncontrolled or significant cardiovascular disease, including any of the following:

  * A myocardial infarction within 6 months
  * Uncontrolled angina within 3 months
  * Congestive heart failure within 3 months
  * Diagnosed or suspected congenital long QT syndrome
  * Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or Torsades de Pointe)
  * Prolonged QTcF interval > 450 msec on pre-entry ECG
* Atypical BCR-ABL1 transcript not quantifiable by RQ-PCR.
* Another primary malignant disease, which requires systemic treatment (chemotherapy or radiation) Severe and/or life-threatening medical disease including acute liver disease
* History of significant congenital or acquired bleeding disorder unrelated to cancer
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of dasatinib
* Patients actively receiving therapy with strong CYP3A4 inhibitors and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug
* Patients who are currently receiving treatment with any medications that have the potential to prolong the QT interval and the treatment cannot be either discontinued or switched to a different medication prior to starting study drug
* Female patients who are: pregnant, breast feeding or potentially fertile without a negative pregnancy test prior to baseline or unwilling to use contraception on trial
* Previous history of pericarditis or pleuritis
* History of non-compliance, abuse of alcohol, illicit drugs, severe psychiatric disorders or other inability to grant informed consent.
* Current treatment for depression.
* Hypersensitivity to any interferon preparation;
* Autoimmune hepatitis or a history of autoimmune disease;
* Pre-existing thyroid disease unless it can be controlled with conventional treatment;
* Epilepsy and/or compromised central nervous system (CNS) function;
* HCV/HIV patients

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
major molecular response rates | 1 year
  defined as ≤0.1% BCR-ABL1 on the MMR International Scale

SECONDARY OUTCOMES:
overall survival | 2 years
quality of life | up to 18 months (after 3, 6, 12, 18 months)
Rate of CCgR | up to 18 months (after 3, 6, 12 and 18 months)
Rate of MR4.0 and MR4.5 | up to 24 months (after 3, 6, 12, 15, 18, and 24 months)

CONTACTS AND LOCATIONS:
Overall Officials: Henrik Hjorth-Hansen, MD PhD, Study Chair — Norwegian University of Science and Technology
Locations (14):
- Helsinki University Central Hospital, Helsinki, Finland
- Norway (5):
  - Bergen University Central Hospital, Bergen
  - Rikshospitalet, Oslo
  - Stavanger University Hospital, Stavanger
  - University Hospital of Northern Norway, Tromsø
  - St Olavs Hospital - Trondheim University Hospital, Trondheim
- Sweden (8):
  - Linköping University Hospital, Linköping
  - Sunderby Sjukhus, Luleå
  - Lund University Hospital, Lund
  - Örebro University Hospital, Örebro
  - Karolinska University Hospital, Stockholm
  - Sundsvall County Hospital, Sundsvall
  - Umeå University Hospital, Umeå
  - Uppsala University Hospital, Uppsala

REFERENCES:
- [Result] Hjorth-Hansen H, Stentoft J, Richter J, Koskenvesa P, Hoglund M, Dreimane A, Porkka K, Gedde-Dahl T, Gjertsen BT, Gruber FX, Stenke L, Eriksson KM, Markevarn B, Lubking A, Vestergaard H, Udby L, Bjerrum OW, Persson I, Mustjoki S, Olsson-Stromberg U. Safety and efficacy of the combination of pegylated interferon-alpha2b and dasatinib in newly diagnosed chronic-phase chronic myeloid leukemia patients. Leukemia. 2016 Sep;30(9):1853-60. doi: 10.1038/leu.2016.121. Epub 2016 May 2. PMID 27133821
- [Derived] Huuhtanen J, Ilander M, Yadav B, Dufva OM, Lahteenmaki H, Kasanen T, Klievink J, Olsson-Stromberg U, Stentoft J, Richter J, Koskenvesa P, Hoglund M, Soderlund S, Dreimane A, Porkka K, Gedde-Dahl T, Gjertsen BT, Stenke L, Myhr-Eriksson K, Markevarn B, Lubking A, Dimitrijevic A, Udby L, Bjerrum OW, Hjorth-Hansen H, Mustjoki S. IFN-alpha with dasatinib broadens the immune repertoire in patients with chronic-phase chronic myeloid leukemia. J Clin Invest. 2022 Sep 1;132(17):e152585. doi: 10.1172/JCI152585. PMID 36047494